CLINICAL TRIAL: NCT05223790
Title: Assessment of the NIPE in Very Premature Infant Ventilated and Sedated in Neonatal Reanimation.
Acronym: NIPEpréma
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0238
Record Dates: First submitted 2021-12-17; First posted 2022-02-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Neonatal; Pain Measurement; Reanimation
Keywords: NIPE; Newborn Infant Parasympathetic Evaluation; Pain measurement; Neonatal care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pain measurement during care procedures in neonatal reanimation — Pain measurement during care procedures in neonatal reanimation

SUMMARY:
The Newborn Infant Parasympathetic Evaluation (NIPE) was developed as a method of analysis of the heart rate variability. The monitor gives a value between 0 (low value of the parasympathetic component) and 100 (high value of the parasympathetic component).

So far, the measure of the heart failure variability by using the NIPE in infant born very premature ventilated and sedated in neonatal reanimation has not been realised and validated as an evaluation method of the pain and discomfort related to neonatal care.

ELIGIBILITY:
Inclusion Criteria:

* Infant born very premature before 34 weeks of amenorrhoea + 0 day
* Age ≤ 7 days
* Admitted in neonatal reanimation
* Sedated, intubated, ventilated

Exclusion Criteria:

* High frequency oscillation ventilation
* Heart rate non sinusal
* Inotropes and atropine
* Opposition from the guardian of parental authority
* Difficulty of comprehension or communication making the parental information impossible

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant born very premature and aged less than 8 days ventilated and sedated in neonatal reanimation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Variation of the NIPE measures between before and during care. | From 10 minutes before the care to 10 minutes after the beginning of the care
  Average of NIPE mesures 10 minutes before the begining of the care and 10 minutes after.

SECONDARY OUTCOMES:
Correlation between the variation of the NIPE measures and the variation of PIPP-R behavioural scale between each period | From 10 minutes after the beginning of the care to 10 minutes after the end of the care
  The average of NIPE mesures 10 minutes before care, 10 minutes after the begining and 10 minutes after the end of the care were collected. And the same for the PIPP-R behavioral scale mesures.
Correlation between the NIPEmin and the PIPP-R behavioural scale for each period | From 10 minutes before the care to 10 minutes after the care
  The lowest NIPE mesures during the 10 minutes before care, 10 minutes after the begining and 10 minutes after the end of the care were collected. And the same for the PIPP-R behavioral scale mesures.
The discriminant power of the NIPE to split the painful population and the non-painful population determined by a threshold at 6 on the PIPP-R scale | From 10 minutes before the care to 10 minutes after the care
  Study the discriminant power of the NIPE to split the painful population and the non-painful population determined by a threshold at 6 on the PIPP-R scale

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukris, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France